CLINICAL TRIAL: NCT02479503
Title: Antibiotic Prophylaxis in Adult Heart Transplantation: a French National Survey
Acronym: ATC
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: ATC
Record Dates: First submitted 2015-06-12; First posted 2015-06-24 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2015-06

CONDITIONS: Antibiotic Prophylaxis; Adult Heart Transplantation
Keywords: antibiotic prophylaxis heart transplantation
MeSH Terms: interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- French Adult Heart Transplantation Center: All center performing adult heart transplantation in France in 2015.
  Interventions: Procedure: Antibiotic prophylaxis in adult heart transplantation

INTERVENTIONS:
Procedure: Antibiotic prophylaxis in adult heart transplantation

SUMMARY:
The study focuses on the antibiotic prophylaxis use in adult heart transplantation in France.

DETAILED DESCRIPTION:
In adult heart transplantation, clinical situations differ between patients (elective, emergency, redux surgery, ventricular assisting device or extracorporeal live saving). At investigator's knowledge, there is not recommendations in France about antibiotic prophylaxis in adult heart transplantation. So, investigators aimed to study the antibiotic prophylaxis use in adult heart transplantation in France.

Investigators conduct a French national survey about antibiotic prophylaxis used in adult heart transplantation center. Clinical situations such as elective, emergency, redux surgery, ventricular assisting device or extracorporeal live saving are investigated.

Study was performed after Institutional approval was obtained from the local Ethics Committee (Comite de Protection des Personnes Nord Ouest III). An electronic survey was sent to all French adult heart transplantation centers (22) on march 1st, 2015. Reminders were planned on week 2 and 4 after initial sending. On june 2015, nonresponding centers were contacted by phone. Data were collected by a single investigator.

ELIGIBILITY:
Inclusion Criteria:

* All French centers performing adult heart transplantation in 2015

Exclusion Criteria:

* not responding center
* no adult heart transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All French centers perfoming adult heart transplantation in 2015.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Class of antibiotic used as prophylaxis in adult heart transplantation | one year

SECONDARY OUTCOMES:
Class of antibiotic used as prophylaxis in adult heart transplantation in regard to clinical situation | one year
  elective, emergency, redux surgery, ventricular assisting device or extracorporeal live saving
Fungal prophylaxis in adult heart transplantation | one year
Other prophylactic measures (isolation, specific room, family visits) used in adult heart transplantation | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, Normandy, France

REFERENCES:
- [Background] Zuckermann A, Barten MJ. Surgical wound complications after heart transplantation. Transpl Int. 2011 Jul;24(7):627-36. doi: 10.1111/j.1432-2277.2011.01247.x. Epub 2011 Mar 21. PMID 21418335
- [Background] Montoya JG, Giraldo LF, Efron B, Stinson EB, Gamberg P, Hunt S, Giannetti N, Miller J, Remington JS. Infectious complications among 620 consecutive heart transplant patients at Stanford University Medical Center. Clin Infect Dis. 2001 Sep 1;33(5):629-40. doi: 10.1086/322733. Epub 2001 Aug 6. PMID 11486285
- [Background] Ramos A, Asensio A, Munez E, Torre-Cisneros J, Blanes M, Carratala J, Segovia J, Munoz P, Cisneros JM, Bou G, Aguado JM, Cervera C, Gurgui MM. Incisional surgical infection in heart transplantation. Transpl Infect Dis. 2008 Jul;10(4):298-302. doi: 10.1111/j.1399-3062.2008.00316.x. Epub 2008 May 15. PMID 18482203